CLINICAL TRIAL: NCT04523753
Title: Emergency Endoscopy for Gastrointestinal Bleeding Situations in Surgical Patients
Brief Title: Endoscopy for Bleeding Situations in Surgical Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: Olena
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-06

CONDITIONS: Hemorrhage
Keywords: surgical patients, gastrointestinal bleeding
MeSH Terms: conditions — Hemorrhage; Gastrointestinal Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: emergency endoscopy — emergency endoscopy for gastrointestinal bleeding situation before or after surgery

SUMMARY:
Retrospective analysis of surgical patients with relevant gastrointestinal bleeding situations and indication for endoscopy for bleeding

DETAILED DESCRIPTION:
We performed an analysis of all adult, surgial patients with indication for emergency endoscopy because of relevant gastrointestinal bleeding situations. A retrospective analysisof the incidence, causes, endoscopic findings and therapy and the outcome of bleeding situations during a 24-mounths interval in the years 2017, 2018 and 2019 was performed at our tertiary centre. Informed consent was obtained from all participants. Patient records as well as database were analyzed for therapy-specific items.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the University Hospital of Tübingen Department of General, Visceral and Transplantation Surgery with gastrointestinal bleeding situations

Exclusion Criteria:

* younger patients
* patients without indication for emergency endoscopy for bleeding situations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of the University Hospital of Tübingen Department of General, Visceral and Transplantation Surgery with gastrointestinal bleeding situations were enrolled for this retrospective analysis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
rate identification of bleeding sources | 24 months
  endoscopic reports with identification of bleeding sources

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No